CLINICAL TRIAL: NCT00414037
Title: Subchronic Effects of Eszopiclone (Lunesta) on Pain Behavior and Circuitry in Primary Insomnia
Brief Title: How do Sleeping Pills Affect Pain in the Brain?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding terminated by sponsor, insufficient data collection
Sponsor: University of California, San Diego (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Martin Paulus, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 060881
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Primary Insomnia
Keywords: insomnia; lunesta; eszopiclone; pain; fMRI
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eszopiclone (Lunesta) 3mg (Experimental): Subchronic (1-week) administration of 3mg Lunesta (eszopiclone)
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): Placebo-treated group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone
  Arms: eszopiclone (Lunesta) 3mg
Drug: Placebo — Placebo-treatment
  Arms: Placebo

SUMMARY:
If you are age 20-55 years old and have trouble falling or staying asleep, then please contact a UCSD research team to find out how a study drug affects these symptoms and how your brain works. This is a one-week experimental pain research study using a study drug compared to placebo. Your participation will include questionnaires, a physical exam and functional Magnetic Resonance Imaging (fMRI) brain imaging techniques. We will test pain perception by applying brief mild to moderate heat pain to the forearm, and also have you perform simple computer tasks while we image and record brain activity using fMRI.

DETAILED DESCRIPTION:
It is well known that chronic pain syndromes are associated with alterations in sleep continuity and sleep architecture. Similarly, recent evidence indicates that sleep deprivation interferes with normal pain perception producing hyperalgesic changes, and with the regular analgesic effects of certain pain drugs (reviewed in Kundermann B et al., 2004). However, the role of the nonbenzodiazepine hypnotic agents in pain perception is not well understood. Lunesta (eszopiclone), unlike other nonbenzodiazepine sleep medications, is approved for long-term use (no significant addictive effects of the drug are observed following the treatment of up to 6mo). Its antinociceptive properties have not been examined and, if found, could potentiate the use of this drug for pain control, especially in patients with comorbid chronic pain and insomnia.

The objective of this proposal is to use Functional Magnetic Resonance Imaging (fMRI) with an experimental pain paradigm in a group of chronic insomnia patients. The study will consist of three sessions, the first of which will include questionnaires, and a mental and physical health evaluation including an EKG and blood draw. Following the initial screening session subjects will be randomly assigned to either the study drug or placebo groups, and complete 2 additional identical study sessions using fMRI. The first fMRI session will be before taking the drug/placebo, and the second session will be after taking the study drug/placebo nightly for 1 week. During these fMRI sessions, subjects will undergo psychophysical testing of their sensitivity to warmth and heat and will rate various temperatures for pain intensity and pain unpleasantness. Subjects will also complete additional tasks including motor inhibition and face matching during scanning.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55
* Primary Insomnia

Exclusion Criteria:

* Certain medical conditions/medications
* MRI related

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sleep and pain ratings following 1 week of treatment as compared to baseline | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Department of Psychiatry, Laboratory of Biological Dynamics and Theoretical Medicine, La Jolla, California, United States